CLINICAL TRIAL: NCT04910659
Title: Effectiveness of Acupuncture in Prevention of Postoperative Sore Throat Due to Classical Laryngeal Mask
Brief Title: Acupuncture in Prevention of Postoperative Sore Throat Due to Classical Laryngeal Mask
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: E1-19-124
Record Dates: First submitted 2021-03-30; First posted 2021-06-02 (Actual); Last update posted 2021-06-08 (Actual); Status verified 2021-03

CONDITIONS: Acupuncture; Laryngeal Mask Airway; Pain, Postoperative; Sore Throat
Keywords: Sore Throat; Laryngeal Mask Airway; Acupuncture
MeSH Terms: conditions — Pain, Postoperative; Pharyngitis | interventions — Acupuncture Therapy

STUDY DESIGN:
Intervention Model Description: prospective randomized controlled study
Who Masked: Participant, Outcomes Assessor
Masking Description: double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- acupuncture (Active Comparator): Group1, laser acupuncture was applied to each of the previously described P6, LI4 and LI 11 points on both arms with laser acupuncture device (Sedatelec Premio 32) for 30 seconds
  Interventions: Other: acupuncture
- false acupuncture (Sham Comparator): P6, LI4 and LI 11 points on both arms with laser acupuncture device (Sedatelec Premio 32) for 30 seconds while laser acupuncture closed
  Interventions: Other: acupuncture

INTERVENTIONS:
Other: acupuncture — P6, LI4 and LI 11 stimulation

SUMMARY:
the aim of our study is to investigate if stimulation of the P6, LI4 and LI11 acupuncture points via laser acupuncture prevents sore throat caused by the classic laryngeal mask.

DETAILED DESCRIPTION:
Our study is planned as a prospective, randomized, controlled, single blind. The details of the study are explained to the patients and their written informed consents are obtained.

Using the randomization program, the patients are divided into group 1 (acupuncture group) and group 2 (control group). Preoxygenation (100% oxygen with balloon and mask for 3 minutes) and midozolam 0.02 mg / kg and fentanyl 2 mcgr / kg are administered to both groups. In Group1, laser acupuncture is applied to each of the previously described P6, LI4 and LI 11 points on both arms with laser acupuncture device (Sedatelec Premio 32) for 30 seconds. In Group 2, same procedure is performed for 30 seconds while laser acupuncture closed. Then, propofol 2mg / kg is administered and a laryngeal mask is placed after 90 seconds in both groups. Maintenance anesthesia is provided with sevofurane and remifentanil infusion.

ELIGIBILITY:
Inclusion Criteria:

* Patients who recieved general anesthesia with LMA
* surgery duration < 2 hours
* between 18-60 years of age
* ASA1-2 scores

Exclusion Criteria:

1. Being younger than 18 years old or being over the age of 60
2. Patients with an ASA score of 3 and greater than 3
3. Active infections in the area to be acupuncture.
4. Prolonged bleeding time
5. Liver failure
6. Renal insufficiency
7. Pregnancy
8. Heart failure 9 . Patients less than 30 kg

10. Uncontrolled hypertension

11. Uncontrolled diabetes, pheochrocytoma, thyroid dysfunction

12. Those who do not have the ability to read and sign the consent form

13. Patients with gastroesophageal reflux

14. History of any herbal medicine use

15. Patients who do not want to sign the consent form

16. Patients with difficult LMA placement

17.Patients who cannot have LMA placement at one time

18. Intubated patients in whom LMA could not be placed

19 Patients whose operation time exceeds two hours

20 .Patients whose operation time is less than 30 minutes

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-07-15 (Estimated); Study Completion 2021-07-30 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline sore throat at 24 h | baseline to 24 hours
  postoperative sore throat is evaluated at 0th, 2th, 6th, 12th, 24th hours with using no, mild, moderate, severe scale.
Change from Baseline postoperative cough at 24 hours | baseline to 24 hours
  postoperative cough is evaluated at 0th, 2th, 6th, 12th, 24th hours and recorded as present or absent
Change from Baseline postoperative snoring at 24 hours | baseline to 24 hours
  postoperative snoring is evaluated at 0th, 2th, 6th, 12th, 24th hours and recorded as present or absent

SECONDARY OUTCOMES:
duration of operation | 24 hour
resistance to Laringeal mask placement (none, mild, moderate, severe) | 24 hours
  1. none
  2. mild
  3. moderate
  4. severe
time taken for Laringeal mask placement (opening of the mouth for placement and time to confirmation of LMA placement with capnograph and auscultation | 24 hours
  time from opening of the mouth for placement to confirmation of LMA placement with capnograph and auscultation

CONTACTS AND LOCATIONS:
Overall Officials: FERYAL AKÇAY, Principal Investigator — Ankara City Hospital Bilkent; FERYAL AKÇAY, Study Chair — Ankara City Hospital Bilkent
Locations (1):
- Ankara City Hospital Bilkent, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided